CLINICAL TRIAL: NCT01726816
Title: A Phase II, Multicenter, Randomized, Double Blind, Double-dummy, 16-week, Placebo Controlled Study to Evaluate the Efficacy and Safety of Probucol in Patients With Nephropathy Due to Type 2 Diabetes.
Brief Title: Efficacy and Safety Study of Probucol in Patients With Diabetic Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 009-KOA-1201i
Record Dates: First submitted 2012-10-31; First posted 2012-11-15 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetic nephropathy; Albumin creatinine ratio; Probucol
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Probucol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Probucol 250mg/day (Experimental): Probucol 250mg group: probucol 250mg 2 tablets, 16 weeks
  Interventions: Drug: Probucol 250mg/day
- Probucol 500mg/day (Experimental): Probucol 500mg group: probucol 250mg 2 tablets, 16 weeks
  Interventions: Drug: Probucol 500mg/day
- Placebo (Placebo Comparator): Placebo group: placebo 2 tablets, 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Probucol 250mg/day — Probucol 250mg + Placebo
  Other Names: Probucol 250mg group: probucol 250mg 2 tablets, 16 weeks
  Arms: Probucol 250mg/day
Drug: Probucol 500mg/day — Probucol 500mg + Placebo
  Other Names: Probucol 500mg group: probucol 250mg 2 tablets, 16 weeks
  Arms: Probucol 500mg/day
Drug: Placebo — Probucol matching placebo
  Other Names: placebo 2 tablets, 16 weeks
  Arms: Placebo

SUMMARY:
This trial is randomized, placebo-controlled, double blind, double dummy, multi-centre trial.

* Screening period (4 week)
* Double blind treatment period (16 weeks)

DETAILED DESCRIPTION:
1. Usage: 16 week, BID, Prescribed Oral with the breakfast and dinner
2. Dosage:Placebo group: placebo 2 tablets, 16 weeks Probucol 250mg group: probucol 125mg 2 tablets, 16 weeks Probucol 500mg group: probucol 250 mg 2 tablets, 16 weeks

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female diagnosed with type 2 diabetes mellitus and must be aged 20 to 75 years at the time of screening visit
2. Urinary albumin excretion > 300 mg/g Cr at screening visit
3. Subjects administered ACEI or ARB without changing dosage prior to 3 months at the screening visit (if subjects administered ACEI or ARB)
4. Subjects administered statins without changing dosage prior to 3 months at the screening visit(if subjects administered statins) or subjects have no plan to administered to statin(if subjects is not administered statin)
5. 15 mL/min ≤ eGFR ≤ 90 mL min
6. Subjects must be willing and able to give signed and dated written informed consent.

Exclusion Criteria:

1. Type 1 DM or gestational diabetes
2. Subjects on Renal replacement therapy or Renal transplantation prior to Screening visit
3. Ventricular arrhythmia (multiple and multifocal premature ventricular contractions)
4. Cardiac damage (abnormally levels of Troponin I)
5. Subject with medical history of cardiac syncope or primary syncope
6. Has condition that may prolong QTc interval (for man QTc interval>450msec, for woman QTc interval>470msec) at screening
7. Pregnant or lactating woman before randomization
8. Inflammatory bowel disease (ulcerative colitis, Crohn's disease)
9. Cholestasis
10. Congestive heart failure
11. Subjects with a myocardial infarction, Unstable angina, or cerebral infarction within the latest 6 months
12. Subjects has a diagnosis of NYHA grade III-IV status
13. AST or ALT is 3.0 times higher than the upper limit of the normal range
14. Active hepatitis Or Liver cirrhosis
15. Subjects with Hyperkalemia (K>5.5 mEq/L)
16. Subjects with Renal Artery stenosis
17. Subjects with Malignancy within the 5 years at the time of screening visit(except for treated Basal cells carcinoma or squamous cell carcinoma)
18. Urinary tract disease (urinary tract infection, Neurogenic bladder)
19. Kidney disease (nephritis, chronic glomerulonephritis or polycystic kidney disease)
20. Has an allergic history to probucol
21. HbA1c > 9%
22. Systolic blood pressure ≥ 160 mmHg or Diastolic blood pressure ≥ 100 mmHg
23. Subjects taken probucol within 3 months prior to Screening
24. The subject has received an investigational product or biological agent within 3 months prior to screening
25. Subjects otherwise judged by the investigator or sub investigator to be inappropriate for inclusion in the trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
A/C ratio | 16 week
  The change in the A/C ratio from baseline to the end of treatment(16 week) [Time Frame: baseline to 16 weeks]

SECONDARY OUTCOMES:
Serum creatinine | 16 week
  The change in the Serum creatinine from baseline to the end of treatment.
eGFR | 16 week
  The change in the eGFR from baseline to the end of treatment(16 week)
cystatin C | 16 week
  The change in the cystatin C from baseline to the end of treatment(16 week)
urine albumin | 16 week
  The change in the urine albumin from baseline to the end of treatment(16 week)
P/C ratio | 16 week
  The change in the P/C ratio from baseline to the end of treatment(16 week)

OTHER OUTCOMES:
Total Cholesterol | 16 week
  The change in the Total cholesterol from baseline to the end of treatment(16 week)
Triglyceride | 16 week
  The change in the Triglyceride from baseline to the end of treatment(16 week)
LDL-C | 16 week
  The change in the LDL-C from baseline to the end of treatment(16 week)
HDL-C | 16 week
  The change in the HDL-C from baseline to the end of treatment(16 week)
oxidized LDL | 16 week
  The change in the oxidized LDL from baseline to the end of treatment(16 week)
d-ROM | 16 week
  The change in the d-ROM from baseline to the end of treatment(16 week)
urinary fibronectin | 16 week
  The change in the urinary fibronectin from baseline to the end of treatment(16 week)
urinary transferrin | 16 week
  The change in the urinary transferrin from baseline to the end of treatment(16 week)
insulin | 16 week
  The change in the insulin from baseline to the end of treatment(16 week)
c-peptide | 16 week
  The change in the c-peptide from baseline to the end of treatment(16 week)

CONTACTS AND LOCATIONS:
Overall Officials: MoonKyu Lee, professor, Study Chair — Samsung Medical Center
Locations (16):
- South Korea (16):
  - The Catholic university of Korea, Bucheon St. Mary's Hospital, Bucheon-si
  - Kyungpook National University, Daegu
  - Yeungnam University Medical Center, Daegu
  - Gil Hospital, Incheon
  - Inha University Hospital, Incheon
  - Chonbuk national University Hospital, Jeonju
  - Eulji Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Kangnam Sacred Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyunghee Univ Hospital at Kangdong, Seoul
  - Samsumg Medical Center, Seoul
  - Severance Hospital, Seoul
  - Seoul National University Bundang Hospital, SungNam
  - St. Vincent Hospital, Suwon
  - UIJEONGBU ST. MARY's HOSPITAL, Uijeongbu-si

REFERENCES:
- [Derived] Jin SM, Han KA, Yu JM, Sohn TS, Choi SH, Chung CH, Park IeB, Rhee EJ, Baik SH, Park TS, Lee IK, Ko SH, Hwang YC, Cha BS, Lee HW, Nam MS, Lee MK. Probucol in Albuminuric Type 2 Diabetes Mellitus Patients on Renin-Angiotensin System Blockade: A 16-Week, Randomized, Double-Blind, Placebo-Controlled Trial. Arterioscler Thromb Vasc Biol. 2016 Oct;36(10):2108-14. doi: 10.1161/ATVBAHA.116.308034. Epub 2016 Aug 4. PMID 27493100